CLINICAL TRIAL: NCT05507736
Title: Feasibility and Safety of the Use of Acupuncture in the Prevention of Late-onset Diarrhea Associated With Irinotecan in Pediatric Patients With Solid Tumors: Controlled Pilot Study
Brief Title: Feasibility and Safety of Acupuncture in the Prevention of Late Irinotecan-related Diarrhea in Pediatric Patients
Acronym: AIP2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PS-20-21
Record Dates: First submitted 2022-07-06; First posted 2022-08-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer; Solid Tumor
Keywords: cancer; children; diarrhea; acupuncture; irinotecan
MeSH Terms: conditions — Neoplasms; Diarrhea | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Pre-post feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Pre-Post feasibility treatment On the first cycle of irinotecan, the patient does not receive any intervention, we only collect data. This is the control cycle.
  There will be a single study group that will be used at the same time as your own control. On the second cycle of irinotecan, the patient receives acupuncture. There will be a single study group that will be used at the same time as your own control.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — 13 Indwelling, sterile and disposable needles (SEIRIN NEW PYONEX® from 0.9 mm in length and 0.22 mm in diameter) on day 1 and 5 of the second cycle of irinotecan leaving them inserted for 4 days.
  Other Names: Indwelling, sterile and disposable needles (SEIRIN NEW PYONEX®)

SUMMARY:
To evaluate the feasibility of an acupuncture protocol in the prevention of late diarrhea due to irinotecan in pediatric patients with solid tumors, a pre-post pilot study will be conducted.

Pre-post pilot study non-randomized, open label, single arm study. There will be a single study group that will be used at the same time as your own control. The intervention will take place for approximately one year.

DETAILED DESCRIPTION:
Pre-post pilot study non-randomized, open label, single arm study.

The objective of this pilot study is to demonstrate that cancer acupuncture pediatric treatment is a safe and feasible treatment in the prevention of late-onset diarrhea related to with irinotecan.

This pilot study will include patients between 0 and 18 years of age with a solid tumor (nephroblastoma, neuroblastoma, central nervous system tumors and rhabdomyosarcoma) receiving their first cycle of irinotecan, in our center, at 50 mg/m2/intravenous dose daily for five days (cumulative dose weekly = 250 mg/m2) and who do not receive concomitant abdominal radiotherapy. Acupuncture will be applied as a complementary treatment along with the usual regimen of prophylaxis and treatment of late diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 0 to 18 years old with solid tumors who start treatment in our center with irinotecan at 50 mg/m2/intravenous dose in day hospital.
* Blood tests prior to the start of the appropriate chemotherapy cycle to receive acupuncture with continuous stimulation needle insertion: neutrophils greater or equal to 1000 cells/mm3 and platelets greater than or equal to 50,000 cells/mm3.
* Signature of informed consent by parents in the case of children under 12 years of age and assent of the minor.
* Signature of informed consent in the case of those over 12 years of age

Exclusion Criteria:

* Participate in a clinical trial that is developed in the Pediatric Oncology Area of the Hospital Sant Joan de Deu where acupuncture intervention is not permitted.
* Have received acupuncture treatment in the last ten days.
* Receive concomitant abdominal radiotherapy.
* Have diarrhea on day 1 of the cycle

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity during the procedure | Day 1
  Evaluation of pain intensity during the insertion procedure of the indwelling needles. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the procedure | Day 5
  Evaluation of pain intensity during the insertion procedure of the indwelling needles. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.

SECONDARY OUTCOMES:
Pain intensity during the intervention | Day 1
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 2
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 3
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 4
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 5
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 6
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 7
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 8
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Pain intensity during the intervention | Day 9
  Evaluation of the intensity of the pain during the days that the indwelling needles remain inserted. It will be evaluated with the same tools as the variable major. The scales will be used: crying scale (0-8) (<3 years), Wong-Baker scale of faces for cooperative children (0-10) (>3 years) and numerical scale (0-10) for collaborating children (>6 years). Higher scores mean a worse result.
Side effects | Day 9
  Registry of other local adverse effects of acupuncture. will be delivered families recorded some items on day 9 of the second cycle (intervention cycle): local infection, hematoma, and skin damage.
Degree of severity of diarrhea | Day 1
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 2
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 3
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 4
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 5
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 6
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 7
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 8
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 9
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 10
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 11
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 12
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 13
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Degree of severity of diarrhea | Day 14
  Degree of severity of diarrhea according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (1-5). It will be evaluated after collection of data from the registration tables that families fill out. Higher scores mean a worse result.
  Grade 1: Increase of <4 stools per day over baseline. Grade 2: Increase of 4 - 6 stools per day over baseline Grade 3: Increase of >=7 stools per day over baseline; hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Dose of antidiarrheal drugs | Day 1
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 2
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 3
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 4
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 5
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 6
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 7
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 8
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 9
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 10
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 11
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 12
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 13
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antidiarrheal drugs | Day 14
  Dose of antidiarrheals: the number of daily doses of loperamide (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Prophylactic regimen of cefixime | Day 1
  Prophylactic regimen of cefixime before starting the cycle of irinotecan and the use of regimen prolonged 10 days. (Yes/No)
Abdominal pain treatment-related | Day 1
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 2
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 3
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 4
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 5
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 6
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 7
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 8
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 9
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 10
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 11
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 12
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 13
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Abdominal pain treatment-related | Day 14
  Degree of abdominal pain assessed with a visual analog scale of 0-10. Higher scores mean a worse result.
Satisfaction degree | Day 15
  Degree of satisfaction with acupuncture through a qualitative survey. Three items Yes/No and free comments
Determination of the UGT1A1 polymorphism | Day 1
  Determination of the UGT1A1 polymorphism by blood sample in the analysis of routine performed on day 1 of the first cycle of irinotecan (control cycle).
Nausea | Day 1
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 2
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 3
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 4
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 5
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 6
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 7
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 8
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 9
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 10
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 11
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 12
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 13
  Record whether or not the patient has nausea (YES/NO)
Nausea | Day 14
  Record whether or not the patient has nausea (YES/NO)
Vomiting | Day 1
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 2
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 3
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 4
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 5
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 6
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 7
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 8
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 9
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 10
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 11
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 12
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 13
  Record whether or not the patient has vomiting (YES/NO)
Vomiting | Day 14
  Record whether or not the patient has vomiting (YES/NO)
Dose of antiemetic drugs (ondasentron) | Day 1
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 2
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 3
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 4
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 5
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 6
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 7
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 8
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 9
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 10
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 11
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 12
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 13
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.
Dose of antiemetic drugs (ondasentron) | Day 14
  Dose of antidiarrheals: the number of daily doses of ondasentron (0-4 doses/day) will be recorded. Higher scores mean a worse result.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Martinez, MD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No